CLINICAL TRIAL: NCT01241955
Title: A Temporal Intervention Trial of a CPR Video in the ICU
Brief Title: Temporal Intervention Trial of a CPR Video in the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-P-001820/1
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Admission to ICU
Keywords: CPR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- verbal description of CPR (No Intervention): verbal description of CPR
- Video decision aid (Experimental): Video decision aid of CPR
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid — video of CPR
  Arms: Video decision aid

SUMMARY:
To compare the decision making of family members of patients admitted to the ICU in regards to their CPR preferences for their loved ones with and without the use of a video decision aid.

DETAILED DESCRIPTION:
Surrogate decision makers of patients admitted to an ICU and UNABLE to make decisions for themselves will be asked their choice for CPR preferences for their loved ones. This will occur during the first six months of the study.

After six months, surrogate decision makers of patients admitted to an ICU and unable to make decisions for themselves will view a video decision aid for CPR and then asked their choice for CPR preferences for their loved ones.

ELIGIBILITY:
Inclusion Criteria:

patient admitted to ICU and unable to make decisions with a known surrogate decision maker

Exclusion Criteria:

Cannot speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
CPR preferences | within 48 hours of ICU admission
  CPR preferences for patients admitted to the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States